CLINICAL TRIAL: NCT03602066
Title: A Pilot Phase II Study Evaluating the Role of Chlorine Dioxide on Mucositis for Patients Undergoing Head and Neck Radiotherapy
Brief Title: Study Evaluating The Role of ClO2 on Mucositis for Pt. Undergoing Head/Neck Radiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by pharmaceutical company
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1712123818; NCI-2018-00214 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1712123818 (Other: The University of Arizona Medical Center-University Campus); P30CA023074 (NIH)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — chlorine dioxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (chlorine dioxide sterilization) (Experimental): Patients receive chlorine dioxide sterilization oral rinse over 30 seconds BID from the start of RT to the evening prior to the 1 month RT follow-up appointment.
  Interventions: Drug: Chlorine Dioxide Sterilization; Other: Laboratory Biomarker Analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo oral rinse over 30 seconds BID from the start of RT to the evening prior to the 1 month RT follow-up appointment.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Drug: Chlorine Dioxide Sterilization — Given via oral rinse
  Other Names: Chlorine Dioxide
  Arms: Arm I (chlorine dioxide sterilization)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given via oral rinse
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This pilot randomized phase II trial studies who well chlorine dioxide sterilization works in reducing oral mucositis in patients with stage I-IV head and neck cancer who are undergoing radiotherapy. Chlorine dioxide sterilization may help to treat oral mucositis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate and compare CloSYS Unflavored Oral Rinse effect on the incidence of severe oral oral mucositis (OM) (>= World Health Organization [WHO] grade 3).

SECONDARY OBJECTIVES:

I. To evaluate and compare CloSYS Unflavored Oral Rinse effect on the time to onset of severe OM (>= WHO grade 3).

II. To evaluate and compare CloSYS Unflavored Oral Rinse effect on the duration of severe OM (>= WHO grade 3).

III. To evaluate and compare CloSYS Unflavored Oral Rinse effect in patient reported outcomes as measured by the Oral Mucositis Weekly Questionnaire (OMWQ).

IV. To evaluate and compare CloSYS Unflavored Oral Rinse effect on rates of radiation therapy (RT) interruption.

V. To evaluate and compare CloSYS Unflavored Oral Rinse effect on the oral microbiome.

VI. To evaluate and compare CloSYS Unflavored Oral Rinse effect on salivary TNFalpha, IL-1beta, and IL-6 levels.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM I: Patients receive chlorine dioxide sterilization oral rinse over 30 seconds twice daily (BID) from the start of radiation therapy (RT) to the evening prior to the 1 month RT follow-up appointment.

ARM II: Patients receive placebo oral rinse over 30 seconds BID from the start of RT to the evening prior to the 1 month RT follow-up appointment.

After completion of study, patients are followed up on day 1.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide properly obtained written informed consent
* Pathologically-confirmed diagnosis of head and neck malignancy (stage I-IV)
* Planned to receive high dose RT >= 50 gray (Gy) to visualizable oral cavity and/or oropharyngeal mucosa, with or without administration of concurrent systemic therapy
* Karnofsky performance status of >= 60, within 45 days of registration
* Hematocrit (Hct) > 20 within 90 days of registration to the study
* Normal cognition and willingness to complete OMWQ and Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTAE) forms at each designated time point along with oral rinse diary
* Life expectancy >= 3 months
* Willing to tolerate oral rinsing for 30 second intervals
* Negative serum pregnancy test in females of childbearing age
* Must be willing to use an effective form of birth control if of child bearing potential

Exclusion Criteria:

* Known hypersensitivity to chlorine dioxide products
* Chlorine dioxide product usage within the past 7 days prior to registration for this study
* Utilization of any antibiotic medications (topical or systemic) within past 7 days prior to registration for this study
* Utilization of daily anti-inflammatory or corticosteroid medication (topical or systemic) for chronic indication other than daily low dose aspirin (81 mg)
* Sjogrens disease
* Medically documented glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Baseline hematocrit =< 20%
* Planned daily RT of less than 5 weeks duration
* Known history of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Yi, Principal Investigator — The University of Arizona Medical Center-University Campus
Locations (1):
- The University of Arizona Medical Center-University Campus, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened on 02/14/2019 and 8 subjects were accrued between February 2019 and November 2019. A subject discovered mold in the IP and all IP was returned to manufacturer and the 8 subjects were withdrawn from study. The study closed to accrual and re-opened 01/15/2022. Subjects were recruited from the University of Arizona Cancer Center clinic from 01/15/2022-08/24/2022. The study closed prematurely as the drug manufacturer pulled funding and IP.
  Enrolled = 14
Period: Overall Study
Arm/Group | Arm II (Placebo) | Arm I (Chlorine Dioxide Sterilization)
Started | 8 | 6
Completed | 5 | 6
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Chlorine Dioxide Sterilization) | Arm II (Placebo) | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 61.5 [35 to 75] | 64 [37 to 81] | 61.5 [35 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14
HNC staging [Count of Participants; unit: Participants] — Head and Neck Cancer staging is based on the American Joint Committee on Cancer (AJCC) staging v. 8. Staging is based on the TNM (tumor, lymph node, metastasis) classification. The lower the number, the lower the cancer stage and the better the prognosis for the patient. The higher the stage, the worse the prognosis.
  Participants
    Stage I | 3 | 4 | 7
    Stage II | 0 | 1 | 1
    Stage III | 2 | 2 | 4
    Stage IV | 1 | 1 | 2
Karnofsky Performance Score [Median (Full Range); unit: Score on a scale] — The Karnofsky Performance Status scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities:
  100=Normal no complaints; no evidence of disease; 90=Able to carry on normal activity; minor signs of symptoms of disease; 80=Normal activity with effort; some signs or symptoms of disease; 70=Cares for self; unable to carry on normal activity or do active work; 60=Requires occasional assistance but is able to care for most of his personal needs
  Per the eligibility criteria, the Karnofsky performance score must be >=60
  Score on a scale | 90 [80 to 100] | 90 [80 to 100] | 90 [80 to 100]
Number of teeth [Median (Full Range); unit: teeth] | 22 [2 to 32] | 28.5 [0 to 32] | 25 [0 to 32]
General dental condition [Count of Participants; unit: Participants]
  Fair | 1 | 1 | 2
  Good | 1 | 4 | 5
  Excellent | 4 | 3 | 7
Oral Mucositis (OM) Grade [Count of Participants; unit: Participants] — OM is measured using the WHO scale. 0 (none) = None I (mild) = Oral soreness, erythema II (moderate) = Oral erythema, ulcers, solid diet tolerated III (severe) = Oral ulcers, liquid diet only IV (life threatening) = Oral alimentation impossible
  Participants
    0 (none) | 6 | 7 | 13
    1 (mild) | 0 | 1 | 1
    2 (moderate) | 0 | 0 | 0
    3 (severe) | 0 | 0 | 0
    4 (life-threatening) | 0 | 0 | 0
    Unknown | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Severe Oral Mucositis (OM) (>= World Health Organization [WHO] Mucositis Scale Grade 3)
Description: Will be compared between arms. Analysis will be performed by estimating the proportion with exact 95% binomial confidence interval for each group separately. Statistical testing will use a chi-square test. As an alternative, Fisher?s Exact Test will be used if the minimum expected value is < 5.
  WHO Scale: Grade 0 (none) - None; Grade I (mild) - Oral soreness, erythema; Grade II (moderate) - Oral erythema, ulcers, solid diet tolerated; Grade III (severe) - Oral ulcers, liquid diet only; Grade IV (life-threatening) - Oral alimentation impossible.
  No grade 3 or higher Oral Mucositis was reported on either treatment arm, so no differences were observed.
Time Frame: Up to 30 days post radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Chlorine Dioxide Sterilization) | Arm II (Placebo)
Number analyzed (Participants) | 6 | 8
Participants | 0 | 0

2. Secondary Outcome: Time to Onset of Severe OM (>= World Health Organization [WHO] Mucositis Scale Grade 3)
Description: Will be tabulated and the median week to onset will be computed for each group. Comparison will be performed using a Wilcoxon Rank Sum Test (as the values are unlikely to be normally distributed).
Time Frame: Up to 30 days post radiotherapy
Measure: Median (Full Range); unit: weeks
Arm/Group | Arm I (Chlorine Dioxide Sterilization) | Arm II (Placebo)
Number analyzed (Participants) | 6 | 8
weeks | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Duration of Severe OM (>= World Health Organization [WHO] Mucositis Scale Grade 3)
Description: as for outcome 2
Time Frame: Up to 30 days post radiotherapy
Measure: Median (Full Range); unit: weeks
Arm/Group | Arm I (Chlorine Dioxide Sterilization) | Arm II (Placebo)
Number analyzed (Participants) | 6 | 8
weeks | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Patient Reported Outcomes as Measured by the Oral Mucositis Weekly Questionnaire (OMWQ)
Description: Will be compared between groups using a linear mixed-effects model to account for the correlation among the measurements within an individual.
Time Frame: Up to 30 days post radiotherapy
Population: Due to the limited patient numbers this was not assessed.
Arm/Group | Arm I (Chlorine Dioxide Sterilization) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Rates of Radiotherapy Interruption
Description: Will be tabulated and compared using a chi-square test.
Time Frame: Up to 30 days post radiotherapy
Population: 3 in Arm II did not complete treatment and were not evaluated for treatment interruption
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Chlorine Dioxide Sterilization) | Arm II (Placebo)
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

6. Other Pre Specified Outcome: Oral Microbiome
Description: as for outcome 4
Time Frame: Up to 30 days post radiotherapy
Population: This analysis was not performed due to lack of sufficient sample size.
Arm/Group | Arm I (Chlorine Dioxide Sterilization) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Salivary TNFalpha, IL-1beta, and IL-6 Levels
Description: as for outcome 4
Time Frame: Up to 30 days post radiotherapy
Population: Analysis not performed due to lack of sufficient patient samples.
Arm/Group | Arm I (Chlorine Dioxide Sterilization) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the treatment period. Subjects were seen once per week per standard of care for on-treatment visits. Radiation treatments may be 6 or 7 weeks at the discretion of the treating physician. Vital signs and weight measurement along with grading of common head and neck side effects per common terminology criteria for adverse events (CTCAE v5.0) were performed.
Description: CTCAE items collected include generalized weakness, skin reaction, weight loss, dry mouth, sore throat, dysphagia, anorexia, dysgeusia, voice alteration, and neck edema. These are common adverse events associated with radiation treatments. There were no adverse events related to the chloride dioxide mouthwash.
Arm/Group | Arm I (Chlorine Dioxide Sterilization) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Chlorine Dioxide Sterilization) (N=6) | Arm II (Placebo) (N=8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Chlorine Dioxide Sterilization) (N=6) | Arm II (Placebo) (N=8)
Generalized weakness (General disorders) | 5 (5) | 6 (6)
Weight loss (Investigations) | 6 (6) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 7 (7)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Dysgeusia (Nervous system disorders) | 6 (6) | 7 (7)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Neck edema (General disorders) | 2 (2) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)

LIMITATIONS AND CAVEATS:
This study stopped accrual early as the IP manufacturer terminated the study stopping funding and IP. 14 out of 20 subjects were accrued, 11 of which completed study. Due to early termination with few patients, only the counts of events have been calculated and no testing was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT03602066/Prot_SAP_000.pdf